CLINICAL TRIAL: NCT02330315
Title: Effects of Transcranial Direct Current Stimulation (tDCS) and Transcranial Ultrasound (TUS) on the Perception of Pain and Functional Limitations Due to Osteoarthritis of the Knee.
Brief Title: Effects of tDCS and tUS on Pain Perception in OA of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Highland Instruments, Inc. (Industry)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014P002496
Record Dates: First submitted 2014-12-12; First posted 2015-01-01 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain; Osteoarthritis
Keywords: transcranial direct current stimulation; transcranial ultrasound; non-invasive brain stimulation
MeSH Terms: conditions — Chronic Pain; Osteoarthritis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS + Active TUS (Experimental): Subjects in the experimental group will undergo 20 minutes of active transcranial direct current stimulation (tDCS) and active transcranial ultrasound (TUS).
  Interventions: Device: transcranial direct current stimulation (tDCS); Device: transcranial ultrasound (TUS)
- Sham tDCS + Sham TUS (Sham Comparator): Subjects in the sham group will undergo 20 minutes of sham transcranial direct current stimulation (tDCS) and sham transcranial ultrasound (TUS).
  Interventions: Device: transcranial direct current stimulation (tDCS); Device: transcranial ultrasound (TUS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — Subjects will receive 20 minutes of either active or sham tDCS at intensity of 2mA. The anodal electrode will be placed over the primary motor cortex contralateral to the most painful side, and the cathodal electrode will be placed over the contralateral supraorbital area. In the sham group, the tDCS device will not be active for the full 20 minutes.
Device: transcranial ultrasound (TUS) — Subjects will receive 20 minutes of either active or sham TUS. During active stimulation the ultrasound will be active for the full 20 minutes- however, during sham stimulation the ultrasound will not be active for the full 20 minutes.

SUMMARY:
The purpose of this study is to investigate the effects of transcranial direct current stimulation (tDCS) in conjunction with transcranial ultrasound (TUS) on pain perception and functional limitations in people with osteoarthritis of the knee. The investigators hypothesize that there will be a decrease in pain levels with active stimulation, when compared to sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent to participate in the study.
2. Subjects between 18-85 years old.
3. Diagnosis of chronic osteoarthritis with pain of either the knee as self-reported.

   Prior to beginning baseline procedures this must be confirmed by medical records or a letter from the subject's physician. This document may either be brought in by the subject or retrieved by study staff after a medical release form is signed by the subject. After consent, if the subject fails to provide the necessary documentation or it cannot be retrieved by study staff the subject will be considered a screen fail.
4. Existing knee pain in the past 6 months of at least 3 on a 0-10 VAS scale on average.
5. Pain resistant to common analgesics and medications for chronic pain used as initial pain management such as Tylenol, Aspirin, Ibuprofen, Soma, Parafon Forte DCS, Zanaflex, and Codeine.
6. Having the ability to feel pain as self-reported

Exclusion Criteria:

1. Pregnancy or trying to become pregnant in the next 6 months.
2. History of alcohol or drug abuse within the past 6 months as self-reported.
3. Contraindications to transcranial brain stimulation or TUS, i.e. implanted brain medical devices or implanted brain metallic devices.
4. Unstable medical conditions (e.g. uncontrolled diabetes, uncompensated cardiac issues, heart failure or chronic obstructive pulmonary disease).
5. Epilepsy.
6. Use of carbamazepine within the past 6 months as self-reported.
7. Suffering from severe depression (with a score of >30 in the Beck Depression Inventory)
8. History of unexplained fainting spells as self-reported.
9. Head injury resulting in more than a momentary loss of consciousness
10. History of neurosurgery as self-reported.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Scale | Measured for approximately 2 months
  Changes in the Visual Analogue Scale (VAS) for pain will be measured in order to determine whether anodal transcranial direct current stimulation in conjunction with transcranial ultrasound (applied in a diagnostic mode) is effective in reducing pain in subjects with osteoarthritis knee pain. The investigators will also look at changes in the Von Frey assessment and pain pressure threshold (PPT).

SECONDARY OUTCOMES:
Changes in Mood | Measured for approximately 2 months
  The investigators will measure safety of tDCS and TUS by measuring changes in the Visual Analog Mood Scale (VAMS).
Changes in cognition, attention, and focus | Measured for approximately 2 months
  The investigators will monitor the safety of tDCS and TUS in subjects by measuring any changes in cognition, attention, and focus with the California Computerized Assessment Package (CalCap) mini.
Adverse Events | Measured for approximately 2 months
  At each session, subjects will complete a questionnaire to evaluate potential adverse effects of stimulation (headache, neck pain, mood alterations, and seizures) on a 5-point scale. The scale will also be administered at the follow-ups.
Physical Examinations | Measured for approximately 2 months
  Trained study staff will perform standard physical examinations at several points throughout the study to ensure subject safety. Baseline findings will be compared to the findings observed at the various time points throughout the study to ensure there are no significant changes that may be study related.
Single Leg Standing Balance Test | Measured for approximately 2 months
  The investigators will measure how long the subject can stand on one foot in order to measure any changes in balance
Knee Proprioceptive Test | Measured for approximately 2 months
  Proprioceptive acuity will be assessed by the ability to reproduce passive positioning of the leg with eyes closed.
Knee Extensor/Flexor Force Test | Measured for approximately 2 months
  The investigators will measure whether there are changes in knee extension/flexion abilities.
Knee Range of Motion (ROM) | Measured for approximately 2 months
  The knee range of motion (flexion/extension angle) will be recorded with an electrogoniometer and motion analysis capture system.
Step Test | Measured for approximately 2 months
  Subject will be asked to stand unsupported with the feet parallel to each other and a block 5 cm directly in front of them. Subject will then be advised which leg is the stepping leg and asked to place the whole foot onto the block, then return it fully down to the floor. This procedure will be repeated as fast as possible.
Functional Reach Test | Measured for approximately 2 months
  The investigators will measure changes in subjects ability to complete the functional reach test across the duration of study.
Timed Up and Go Test | Measured for approximately 2 months
  The investigators will measure if there are changes in the walking speed of the subject from the beginning of the study to the end.
Changes in quality of life | Measured for approximately 2 months
  The investigators will use the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) to assess changes in quality of life and physical functioning.
Neurological Examinations | Measured for approximately 2 months
  Trained study staff will perform standard neurological examinations at several points throughout the study to ensure subject safety. Baseline findings will be compared to the findings observed at the various time points throughout the study to ensure there are no significant changes that may be study related.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wagner, PhD, Principal Investigator — Highland Instruments, Inc.
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States